CLINICAL TRIAL: NCT03531294
Title: Intravitreal Aflibercept as Indicated by Real-Time Objective Imaging to Achieve Diabetic Retinopathy Improvement
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Greater Houston Retina Research (Other)
Collaborators: Regeneron Pharmaceuticals (Industry); The Cleveland Clinic (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PRIME
Record Dates: First submitted 2018-04-25; First posted 2018-05-21 (Actual); Last update posted 2021-05-21 (Actual); Status verified 2021-05

CONDITIONS: Diabetic Retinopathy
MeSH Terms: conditions — Diabetic Retinopathy | interventions — aflibercept

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Group 1 (Experimental): Treatment based on central reading center reading evaluation of DRSS (diabetic retinopathy severity scale) level based on OPTOS funds photos.
  Interventions: Drug: Aflibercept Injection
- Group 2 (Experimental): Treatment based on central reading center reading evaluation of DRSS (diabetic retinopathy severity scale) level based leakage index of OPTOS wide field fluorescein angiography.
  Interventions: Drug: Aflibercept Injection

INTERVENTIONS:
Drug: Aflibercept Injection — intravitreal 2mg aflibercept injection
  Other Names: Eyela

SUMMARY:
The PRIME trial will assess the safety of 2 mg intravitreal aflibercept injections (IAI) to achieve and maintain DRSS improvements (2 or more steps) in patients with a baseline DRSS level of 47A to 71A inclusive through 104 weeks as determined by reading center determined DRSS gradings on OPTOS fundus photos and leakage index on OPTOS WF-FA.

DETAILED DESCRIPTION:
Study eyes will be assigned randomly (1:1 ratio) to one of the following 2 treatment arms. Randomization of PDR subjects will be limited to 50% of each arm.

Group 1

Year 1 Subjects will be seen every month, 28 days (+ 7 days), for 52 weeks. All subjects will receive IAI at baseline, after eligibility is confirmed. Week 4 through week 48, subjects will be seen monthly and treated with IAI PRN (pro re nata) according to, same day, central reading center (CRC) determined DRSS level. Monthly treatment with IAI will continue until a greater than or equal to 2 step DRSS level improvement is achieved, relative to screening/baseline DRSS based on CRC assessment OPTOS fundus photos (FP). Subjects who have baseline proliferative diabetic retinopathy (PDR) (DRSS Level 61-71) will continue to receive monthly IAI until a greater than or equal to 2 step DRSS improvement is achieved as determined by CRC assessment of OPTOS fundus photos relative to screening/baseline DRSS, and PDR is quiescent according to the treating investigator. Treatment with IAI will be reinitiated if a 1 step worsening of DRSS occurs compared to best DRSS score achieved, determined by CRC evaluation of OPTOS fundus photos. If such worsening is detected, the subject would resume monthly IAI until best DRSS score or greater is achieved, as determined by CRC assessment of OPTOS fundus photos. In addition, retreatment will also be re-started if new onset neovascularization is identified and is continued until the PDR is quiescent according to the treating investigator.

Year 2 Beginning in year 2 (week 52) subjects will be seen every 56 days (+ 14 days) and treated with IAI PRN (pro re nata) utilizing the same criteria from year 1. All subjects will have a mandatory week 104 visit, where treatment will not be given.

Group 2

Year 1 Subjects will be seen every month, 28 days (+ 7 days), for 52 weeks. All subjects will receive IAI at baseline, after eligibility is confirmed. Week 4 through week 48, subjects will be seen monthly and treated with IAI PRN (pro re nata) according to, same day, CRC determination of DRSS initially, and subsequently of leakage index.

Monthly treatment with IAI will continue until a greater than or equal to 2 step DRSS level improvement is achieved, relative to screening/baseline DRSS based on CRC assessment OPTOS fundus photos (FP). Subjects who have baseline proliferative diabetic retinopathy (PDR) (DRSS Level 61-71) will continue to receive monthly IAI until a greater than or equal to 2 step DRSS improvement is achieved as determined by CRC assessment of OPTOS fundus photos relative to screening/baseline DRSS, and PDR is quiescent according to the treating investigator.

Leakage index as determined by CRC assessment of OPTOS WF-FA at the visit at which a greater than or equal to 2 step DRSS level improvement is achieved will be considered the threshold. Treatment with IAI will be reinitiated if the leakage index increases to 33% above the individual subject threshold leakage index level as determined by CRC evaluation of OPTOS WF-FA. If such worsening is detected, the subject would resume monthly IAI until the threshold leakage index as determined by CRC assessment of OPTOS WF-FA is reached. In addition, retreatment will also be re-started if new onset neovascularization is identified and is continued until the PDR is quiescent according to the treating investigator.

Year 2 Beginning in year 2 (week 52) subjects will be seen every 56 days (+ 14 days) and treated with IAI PRN (pro re nata) utilizing the same criteria from year 1. All subjects will have a mandatory week 104 visit, where treatment will not be given.

If images of insufficient quality are unable to be obtained, in Group 1 or Group 2, subjects will undergo treatment with IAI at principal investigators discretion or designee.

Subjects can have both eyes in the study, if eligibility is met. If both eyes are eligible, one eye will be randomized to group 1 while the other is randomized to group 2. If only one eye is eligible IAI will be provided for the fellow eye as needed according to the treating investigator.

ELIGIBILITY:
Inclusion Criteria:

1. Men or Women > 18 years of age with type 1 or II diabetes mellitus
2. Diabetic Retinopathy, DRSS Level 47A to 71A, as assessed by CRC (enrollment of PDR levels will be limited to 50% of the total population)
3. BCVA in the study eye better than 20/800

Exclusion Criteria:

1. Any prior systemic anti-VEGF treatment or IVT anti-search vascular endothelial growth factor (VEGF) treatment in the study eye within 24 weeks of screening/baseline
2. Any intravitreal or peribulbar corticosteroids in the study eye within 12 weeks of screening/baseline
3. Any prior treatment with Ozurdex or Iluvien in the study eye
4. SD-OCT central subfield thickness (CST) > 320 µm in the study eye
5. Central DME causing visual acuity loss, in which treatment can not be safely deferred for at least 6 months, in the investigator's judgment
6. Current visually significant vitreous hemorrhage in the study eye. Vitreous hemorrhage is allowed as long as DRSS level is 71A or lower.
7. History of panretinal photocoagulation (PRP) in the study eye
8. History of vitrectomy surgery in the study eye
9. Cataract surgery in the study eye within 8 weeks of screening/baseline
10. Pregnant or breast-feeding women
11. Sexually active men* or women of childbearing potential** who are unwilling to practiceadequate contraception during the study (adequate contraceptive measures include stable use of oral contraceptives or other prescription pharmaceutical contraceptives for 2 or more menstrual cycles prior to screening/baseline; intrauterine device [IUD]; bilateral tubal ligation; vasectomy; condom plus contraceptive sponge, foam, or jelly, or diaphragm plus contraceptive sponge, foam, or jelly).

    * Contraception is not required for men with documented vasectomy.

    ** Postmenopausal women must be amenorrheic for at least 52 weeks in order not to be considered of childbearing potential. Pregnancy testing and contraception are not required for women with documented hysterectomy or tubal ligation.
12. If currently receiving diaylisis, must have started treatment more than 12 weeks prior to screening/baseline
13. Uncontrolled blood pressure (defined as > 190/110 mm Hg systolic/diastolic, while seated)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2018-05-23 (Actual); Primary Completion 2021-04-09 (Actual); Study Completion 2021-04-09 (Actual)

PRIMARY OUTCOMES:
Incidence of Adverse Events for diabetic retinopathy subjects who receive intravitreal Aflibercept | 104 weeks
  Assess the safety of 2 mg intravitreal aflibercept injections (IAI) to achieve and maintain DRSS improvements (2 or more steps) in patients with a baseline DRSS level of 47A to 71A inclusive as determined by reading center determined DRSS gradings on OPTOS fundus photos and leakage index on OPTOS WF-FA

SECONDARY OUTCOMES:
Correlation of DRSS and leakage index | 104 weeks
  Correlation of reading-center determined DRSS level and leakage index to determine change in DR severity
Correlation between Reading Center DRSS Level and Physician determined DR severity | 104 weeks
  Correlation of reading-center determined DRSS level and investigator-determined DR severity level based on ophthalmoscopic fundus examination (Physician determined DR severity level will be based on AAO (American Academy of Ophthalmology) simplified grading system: mild NPDR, moderate NPDR, Severe NPDR, low risk PDR, high risk PDR)
Number of IAI | 104 weeks
  Mean and Median number of IVT aflibercept Injections (with and without IAI given for DME)
Mean number of IAI (NPDR VS PDR) | 104 weeks
  Mean number of IVT aflibercept Injections in eyes with baseline NPDR vs PDR through week 52
ETDRS-BCVA change | 104 weeks
  Mean change in Early Treatment Diabetic Retinopathy Study best corrected visual acuity (ETDRS-BCVA)
Changes in Visual Function | 104 weeks
  Changes in visual function outcomes as measured by National Eye Institute Visual Functioning Questionnaire (NEI-VFQ)
DRSS Change | 104 weeks
  Changes in DRSS
Change in Non-Perfusion | 104 weeks
  Change in area of retinal non-perfusion within the macula and periphery
Change in Vascular Leakage | 104 weeks
  Change in relative area of vascular leakage on wide-field fluorescein angiography
Change in microaneurysms | 104 weeks
  Change in number of microaneurysms, assessed by wide-field fluorescein angiography
Change in CST | 104 weeks
  Mean change in central subfield thickness (CST), as assessed by spectral Domain Optical coherence tomography (SD-OCT)
DME development | 104 weeks
  Percentage of subjects, who develop center-involving diabetic macular edema necessitating treatment compared to baseline
PDR Development | 104 weeks
  Percentage of subjects, who develop a new PDR event compared to baseline
Cytokine Levels | 104 weeks
  Corelation of cytokine levels in aqueous humor samples to clinical and imaging outcomes

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Retina Consultants of Houston/The Medical Center, Houston, Texas
  - Retina Consultants of Houston, The Woodlands, Texas

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ehlers JP, Wang K, Vasanji A, Hu M, Srivastava SK. Automated quantitative characterisation of retinal vascular leakage and microaneurysms in ultra-widefield fluorescein angiography. Br J Ophthalmol. 2017 Jun;101(6):696-699. doi: 10.1136/bjophthalmol-2016-310047. Epub 2017 Apr 21. PMID 28432113
- [Background] Wang K, Srivastava SK, Vasanji A, Hu M, Reese J, Stiegel L, and Ehlers JP. "Quantitative ultrawidefield fluorescein angiography and volumetric optical coherence tomography analysis in the REACT Study: A prospective randomized comparative dosage trial evaluating ranibizumab in bevacizumab-resistant diabetic macular edema." Scientific Poster. ARVO Annual Meeting. Baltimore, MD. May 2017.
- [Background] Ehlers JP. "Peripheral and Macular Retinal Vascular Dynamics in DME and RVO Following Aflibercept Therapy: The PERMEATE Study 6-month Results" Scientific presentation. ASRS Annual Meeting. Boston, MA. August 201
- [Background] Kempen JH, O'Colmain BJ, Leske MC, Haffner SM, Klein R, Moss SE, Taylor HR, Hamman RF; Eye Diseases Prevalence Research Group. The prevalence of diabetic retinopathy among adults in the United States. Arch Ophthalmol. 2004 Apr;122(4):552-63. doi: 10.1001/archopht.122.4.552. PMID 15078674
- [Background] Leasher JL, Bourne RR, Flaxman SR, Jonas JB, Keeffe J, Naidoo K, Pesudovs K, Price H, White RA, Wong TY, Resnikoff S, Taylor HR; Vision Loss Expert Group of the Global Burden of Disease Study. Global Estimates on the Number of People Blind or Visually Impaired by Diabetic Retinopathy: A Meta-analysis From 1990 to 2010. Diabetes Care. 2016 Sep;39(9):1643-9. doi: 10.2337/dc15-2171. PMID 27555623
- [Background] Bourne RR, Stevens GA, White RA, Smith JL, Flaxman SR, Price H, Jonas JB, Keeffe J, Leasher J, Naidoo K, Pesudovs K, Resnikoff S, Taylor HR; Vision Loss Expert Group. Causes of vision loss worldwide, 1990-2010: a systematic analysis. Lancet Glob Health. 2013 Dec;1(6):e339-49. doi: 10.1016/S2214-109X(13)70113-X. Epub 2013 Nov 11. PMID 25104599
- [Background] Early photocoagulation for diabetic retinopathy. ETDRS report number 9. Early Treatment Diabetic Retinopathy Study Research Group. Ophthalmology. 1991 May;98(5 Suppl):766-85. PMID 2062512
- [Background] Photocoagulation treatment of proliferative diabetic retinopathy. Clinical application of Diabetic Retinopathy Study (DRS) findings, DRS Report Number 8. The Diabetic Retinopathy Study Research Group. Ophthalmology. 1981 Jul;88(7):583-600. PMID 7196564
- [Background] Diabetic Retinopathy Clinical Research Network; Elman MJ, Aiello LP, Beck RW, Bressler NM, Bressler SB, Edwards AR, Ferris FL 3rd, Friedman SM, Glassman AR, Miller KM, Scott IU, Stockdale CR, Sun JK. Randomized trial evaluating ranibizumab plus prompt or deferred laser or triamcinolone plus prompt laser for diabetic macular edema. Ophthalmology. 2010 Jun;117(6):1064-1077.e35. doi: 10.1016/j.ophtha.2010.02.031. Epub 2010 Apr 28. PMID 20427088
- [Background] Nguyen QD, Brown DM, Marcus DM, Boyer DS, Patel S, Feiner L, Gibson A, Sy J, Rundle AC, Hopkins JJ, Rubio RG, Ehrlich JS; RISE and RIDE Research Group. Ranibizumab for diabetic macular edema: results from 2 phase III randomized trials: RISE and RIDE. Ophthalmology. 2012 Apr;119(4):789-801. doi: 10.1016/j.ophtha.2011.12.039. Epub 2012 Feb 11. PMID 22330964
- [Background] Korobelnik JF, Do DV, Schmidt-Erfurth U, Boyer DS, Holz FG, Heier JS, Midena E, Kaiser PK, Terasaki H, Marcus DM, Nguyen QD, Jaffe GJ, Slakter JS, Simader C, Soo Y, Schmelter T, Yancopoulos GD, Stahl N, Vitti R, Berliner AJ, Zeitz O, Metzig C, Brown DM. Intravitreal aflibercept for diabetic macular edema. Ophthalmology. 2014 Nov;121(11):2247-54. doi: 10.1016/j.ophtha.2014.05.006. Epub 2014 Jul 8. PMID 25012934
- [Background] Fong DS, Girach A, Boney A. Visual side effects of successful scatter laser photocoagulation surgery for proliferative diabetic retinopathy: a literature review. Retina. 2007 Sep;27(7):816-24. doi: 10.1097/IAE.0b013e318042d32c. PMID 17891003
- [Background] Ferris F. Early photocoagulation in patients with either type I or type II diabetes. Trans Am Ophthalmol Soc. 1996;94:505-37. PMID 8981711
- [Background] Writing Committee for the Diabetic Retinopathy Clinical Research Network; Gross JG, Glassman AR, Jampol LM, Inusah S, Aiello LP, Antoszyk AN, Baker CW, Berger BB, Bressler NM, Browning D, Elman MJ, Ferris FL 3rd, Friedman SM, Marcus DM, Melia M, Stockdale CR, Sun JK, Beck RW. Panretinal Photocoagulation vs Intravitreous Ranibizumab for Proliferative Diabetic Retinopathy: A Randomized Clinical Trial. JAMA. 2015 Nov 24;314(20):2137-2146. doi: 10.1001/jama.2015.15217. PMID 26565927
- [Background] Diabetic Retinopathy Clinical Research Network; Wells JA, Glassman AR, Ayala AR, Jampol LM, Aiello LP, Antoszyk AN, Arnold-Bush B, Baker CW, Bressler NM, Browning DJ, Elman MJ, Ferris FL, Friedman SM, Melia M, Pieramici DJ, Sun JK, Beck RW. Aflibercept, bevacizumab, or ranibizumab for diabetic macular edema. N Engl J Med. 2015 Mar 26;372(13):1193-203. doi: 10.1056/NEJMoa1414264. Epub 2015 Feb 18. PMID 25692915
- [Background] Sivaprasad S, Prevost AT, Vasconcelos JC, Riddell A, Murphy C, Kelly J, Bainbridge J, Tudor-Edwards R, Hopkins D, Hykin P; CLARITY Study Group. Clinical efficacy of intravitreal aflibercept versus panretinal photocoagulation for best corrected visual acuity in patients with proliferative diabetic retinopathy at 52 weeks (CLARITY): a multicentre, single-blinded, randomised, controlled, phase 2b, non-inferiority trial. Lancet. 2017 Jun 3;389(10085):2193-2203. doi: 10.1016/S0140-6736(17)31193-5. Epub 2017 May 7. PMID 28494920
- [Background] Mazhar K, Varma R, Choudhury F, McKean-Cowdin R, Shtir CJ, Azen SP; Los Angeles Latino Eye Study Group. Severity of diabetic retinopathy and health-related quality of life: the Los Angeles Latino Eye Study. Ophthalmology. 2011 Apr;118(4):649-55. doi: 10.1016/j.ophtha.2010.08.003. Epub 2010 Oct 29. PMID 21035872
- [Background] Klein R, Knudtson MD, Lee KE, Gangnon R, Klein BE. The Wisconsin Epidemiologic Study of Diabetic Retinopathy XXIII: the twenty-five-year incidence of macular edema in persons with type 1 diabetes. Ophthalmology. 2009 Mar;116(3):497-503. doi: 10.1016/j.ophtha.2008.10.016. Epub 2009 Jan 22. PMID 19167079
- [Background] Klein R, Klein BE, Moss SE. A population-based study of diabetic retinopathy in insulin-using patients diagnosed before 30 years of age. Diabetes Care. 1985 Sep-Oct;8 Suppl 1:71-6. doi: 10.2337/diacare.8.1.s71. PMID 4053957
- [Background] Fundus photographic risk factors for progression of diabetic retinopathy. ETDRS report number 12. Early Treatment Diabetic Retinopathy Study Research Group. Ophthalmology. 1991 May;98(5 Suppl):823-33. PMID 2062515
- [Background] Klein R, Klein BE, Moss SE. How many steps of progression of diabetic retinopathy are meaningful? The Wisconsin epidemiologic study of diabetic retinopathy. Arch Ophthalmol. 2001 Apr;119(4):547-53. doi: 10.1001/archopht.119.4.547. PMID 11296020
- [Background] Wilkinson CP, Ferris FL 3rd, Klein RE, Lee PP, Agardh CD, Davis M, Dills D, Kampik A, Pararajasegaram R, Verdaguer JT; Global Diabetic Retinopathy Project Group. Proposed international clinical diabetic retinopathy and diabetic macular edema disease severity scales. Ophthalmology. 2003 Sep;110(9):1677-82. doi: 10.1016/S0161-6420(03)00475-5. PMID 13129861
- [Background] Brown DM, Schmidt-Erfurth U, Do DV, Holz FG, Boyer DS, Midena E, Heier JS, Terasaki H, Kaiser PK, Marcus DM, Nguyen QD, Jaffe GJ, Slakter JS, Simader C, Soo Y, Schmelter T, Yancopoulos GD, Stahl N, Vitti R, Berliner AJ, Zeitz O, Metzig C, Korobelnik JF. Intravitreal Aflibercept for Diabetic Macular Edema: 100-Week Results From the VISTA and VIVID Studies. Ophthalmology. 2015 Oct;122(10):2044-52. doi: 10.1016/j.ophtha.2015.06.017. Epub 2015 Jul 18. PMID 26198808
- [Background] Brown DM, Nguyen QD, Marcus DM, Boyer DS, Patel S, Feiner L, Schlottmann PG, Rundle AC, Zhang J, Rubio RG, Adamis AP, Ehrlich JS, Hopkins JJ; RIDE and RISE Research Group. Long-term outcomes of ranibizumab therapy for diabetic macular edema: the 36-month results from two phase III trials: RISE and RIDE. Ophthalmology. 2013 Oct;120(10):2013-22. doi: 10.1016/j.ophtha.2013.02.034. Epub 2013 May 22. PMID 23706949
- [Background] Ip MS, Domalpally A, Hopkins JJ, Wong P, Ehrlich JS. Long-term effects of ranibizumab on diabetic retinopathy severity and progression. Arch Ophthalmol. 2012 Sep;130(9):1145-52. doi: 10.1001/archophthalmol.2012.1043. PMID 22965590
- [Background] Ip MS, Domalpally A, Sun JK, Ehrlich JS. Long-term effects of therapy with ranibizumab on diabetic retinopathy severity and baseline risk factors for worsening retinopathy. Ophthalmology. 2015 Feb;122(2):367-74. doi: 10.1016/j.ophtha.2014.08.048. Epub 2014 Nov 18. PMID 25439595
- [Background] Bressler SB, Liu D, Glassman AR, Blodi BA, Castellarin AA, Jampol LM, Kaufman PL, Melia M, Singh H, Wells JA; Diabetic Retinopathy Clinical Research Network. Change in Diabetic Retinopathy Through 2 Years: Secondary Analysis of a Randomized Clinical Trial Comparing Aflibercept, Bevacizumab, and Ranibizumab. JAMA Ophthalmol. 2017 Jun 1;135(6):558-568. doi: 10.1001/jamaophthalmol.2017.0821. PMID 28448655
- [Background] Wykoff CC, Le RT, Khurana RN, Brown DM, Ou WC, Wang R, Clark WL, Boyer DS; ENDURANCE Study Group. Outcomes With As-Needed Aflibercept and Macular Laser Following the Phase III VISTA DME Trial: ENDURANCE 12-Month Extension Study. Am J Ophthalmol. 2017 Jan;173:56-63. doi: 10.1016/j.ajo.2016.09.029. Epub 2016 Oct 1. PMID 27702624
- [Background] Croft DE, van Hemert J, Wykoff CC, Clifton D, Verhoek M, Fleming A, Brown DM. Precise montaging and metric quantification of retinal surface area from ultra-widefield fundus photography and fluorescein angiography. Ophthalmic Surg Lasers Imaging Retina. 2014 Jul-Aug;45(4):312-7. doi: 10.3928/23258160-20140709-07. PMID 25037013
- [Background] Gulshan V, Peng L, Coram M, Stumpe MC, Wu D, Narayanaswamy A, Venugopalan S, Widner K, Madams T, Cuadros J, Kim R, Raman R, Nelson PC, Mega JL, Webster DR. Development and Validation of a Deep Learning Algorithm for Detection of Diabetic Retinopathy in Retinal Fundus Photographs. JAMA. 2016 Dec 13;316(22):2402-2410. doi: 10.1001/jama.2016.17216. PMID 27898976
- [Derived] Kalra G, Wykoff C, Martin A, Srivastava SK, Reese J, Ehlers JP. Longitudinal Quantitative Ultrawidefield Angiographic Features in Diabetic Retinopathy Treated with Aflibercept from the Intravitreal Aflibercept as Indicated by Real-Time Objective Imaging to Achieve Diabetic Retinopathy Improvement Trial. Ophthalmol Retina. 2024 Feb;8(2):116-125. doi: 10.1016/j.oret.2023.09.004. Epub 2023 Sep 9. PMID 37696393
- See also: World Helath Organization (WHO). Global Report on Diabetes. 2016 — http://apps.who.int/iris/bitstream/10665/204871/1/9789241565257_eng.pdf?ua=1&ua=1
- See also: 2016 America Society of Retina Specialists Preferences and Trends Survey — https://www.asrs.org/content/documents/_asrs-pat-slides-2016-final-sm.pdf